CLINICAL TRIAL: NCT06316453
Title: Prospective Assessment of Atherosclerotic Cardiovascular Disease (ASCVD) Risk in Adults (30 Years and Above) in Pakistan: A Multi-Year Study Investigating Incidence, Validation, and Management Strategies
Brief Title: Prospective Assessment of Atherosclerotic Cardiovascular Disease (ASCVD) Risk
Status: Recruiting | Type: Observational
Sponsor: Advanced Education & Research Center (Other)
Collaborators: University of Karachi (Other); Pakistan Cardiac Society (Heart House) (Unknown)
Responsible Party: Sponsor
Other Study IDs: PARADISE-PK-09-03-2024
Record Dates: First submitted 2024-03-12; First posted 2024-03-18 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Atherosclerotic Cardiovascular Diseases (ASCVD)
Keywords: Prospective; Atherosclerotic Cardiovascular Disease (ASCVD); Risk; Pakistan; Management Strategies
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non pre-existing ASCVD: ASCVD risk in adults will be assessed alongside demographics and clinical history. The study will calculate 10-year, 30-year, and lifetime ASCVD risks, incorporating genetic assessment for Apo B. Personalized management recommendations based on ASCVD risk will be provided, and a six-month follow-up will track ASCVD events.
  Interventions: Other: Evaluating ASCVD risk over 10 and 30 year and lifetime

INTERVENTIONS:
Other: Evaluating ASCVD risk over 10 and 30 year and lifetime — Utilizing validated tools such as the Pooled Cohort Equations (PCE) for 10-year ASCVD risk, the 30-year ASCVD risk prediction tool, and lifetime ASCVD risk categories, participants will undergo a thorough risk assessment. This multi-dimensional approach ensures a nuanced understanding of short and long-term cardiovascular risks. Further, The genetic risk for ApoB will be meticulously assessed by genotyping the APOB rs1042031 variant. Subsequently, the calculation of the genetic risk score (GRS) based on risk alleles will provide personalized insight into genetic predispositions related to ASCVD risk. Moreover, Participants will receive personalized management recommendations derived from the ACC/AHA Cardiovascular Risk Assessment Guidelines. These tailored suggestions may encompass dietary programs, lifestyle modifications, and, when indicated, pharmaceutical therapies like statins, aiming to mitigate identified risks effectively

SUMMARY:
This study aims to conduct a 10-year follow-up to assess ASCVD risk in Pakistan among individuals aged 30 years and above without a known history of ASCVD. The focus will be on evaluating ASCVD risk over this specific 10-year timeframe. The study will also validate risk assessment scores for identifying high-risk individuals and examine the incidence rate of ASCVD events during long-term follow-up.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVD) pose a formidable challenge as the leading cause of premature mortality globally, affecting diverse populations across income societies. The dynamic interplay of sex and age significantly influences the trajectory and prognosis of atherosclerotic cardiovascular diseases (ASCVD). Previously perceived as an ailment predominantly afflicting affluent older men, ASCVD has undergone a transformative shift, emerging as an epidemic impacting the productivity of both young men and women. This resonance is particularly pronounced in communities with varying economic backgrounds, including high-income and low-to-middle-income settings. The far-reaching consequences of premature CVD extend beyond the individual, exerting socioeconomic strains on families and societies, especially in lower-income communities. Recognizing the gravity of this situation, the World Health Organization (WHO) initiated the "25 by 25" campaign, aiming to curtail premature mortality from non-communicable diseases, with over 60% attributed to CVD, by 25% before 2025.

While global data on gender- and age-specific variations in CVD risk factors and outcomes have been extensively documented, the local evidence in Pakistan underscores a crucial research gap. A contemporary ST-elevation acute coronary syndrome (STE-ACS) cohort in Pakistan reveals a noteworthy 12% of premature cases (<40 years). A study by Ullah W et al., comprising 15,106 participants from the Cardiac Registry of Pakistan Catheterization Percutaneous Coronary Intervention, reports 7.4% of patients under 40 years. However, comprehensive local evidence on the incidence of ASCVD among the young population remains scarce.

Current risk assessment guidelines, exemplified by the 2019 ACC/AHA Cardiovascular Risk Assessment Guidelines, predominantly employ race- and sex-specific Pooled Cohort Equations (PCE) for predicting 10-year CVD risk, specifically in adults aged 40 to 75. However, these guidelines need more direct applicability to young adults, who often exhibit a paradox of low 10-year ASCVD predicted risk despite harboring a high lifetime risk profile. Acknowledging this discrepancy, the 2018 AHA/ACC cholesterol guideline advocates for estimating lifetime or 30-year ASCVD risk for individuals under 40.

Transitioning from risk assessment to lipid modulation, mainly focusing on low-density lipoproteins (LDL), unveils a pivotal role in atherogenesis. LDL assumes primary responsibility in cholesterol transport. The strategic modulation of lipid profiles has emerged as a central goal for cardiovascular prevention, concentrated on mitigating cardiovascular risk through targeted reduction of LDL-cholesterol using diverse lipid-lowering agents. Recent attention has shifted towards compounds offering nuanced insights into pro-atherogenic risk, with apolipoproteins playing an essential role in regulating lipoprotein metabolism and garnering significant attention in atherosclerosis.

Among the various apolipoproteins, apolipoprotein B (Apo B) emerges as a crucial component integral to all atherogenic lipids, including very low-density lipoproteins (VLDLs), intermediate-density lipoproteins (IDLs), LDLs, and chylomicrons. Existing literature underscores substantial variability in the lipid composition of Apo B lipoproteins, positioning Apo B as superior to total cholesterol and triglyceride levels in predicting cardiovascular risk. However, the predictive role of Apo B versus LDL-cholesterol remains controversial. While some studies advocate for Apo B as a more precise predictor of cardiovascular risk than LDL-cholesterol and non-high-density lipoprotein cholesterol (non-HDL), a recent extensive study involving over 300,000 patients did not establish the superiority of Apo B over LDL-cholesterol in assessing cardiovascular risk. This divergence in findings is mirrored in the 2021 ESC Guidelines on Cardiovascular Disease Prevention in Clinical Practice. Consequently, a series of comprehensive studies is imperative to delineate the precise role of Apo B as a predictor of cardiovascular diseases (CVDs).

In light of Pakistan's escalating ASCVD burden, early identification and optimal management of modifiable risk factors become imperative for prevention. While conclusive studies are lacking, expert recommendations underscore the utility of "total/absolute CVD risk" assessment in guiding management decisions. This study, utilizing the ASCVD risk score and WHO risk score system, aims to evaluate ASCVD risk in young individuals, categorizing risks into low, intermediate, and high groups to guide tailored interventions, be it lifestyle modifications, non-pharmaceutical management, or pharmaceutical interventions, at each specific stage.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of any gender
* Individuals aged 30 years and above
* The study ensured a diverse representation to encompass a broad spectrum of experiences and risk factors within this age group
* Individuals without pre-existing cardiovascular conditions

Exclusion Criteria:

* Individuals with a confirmed diagnosis of ASCVD
* Confirmed cases of cancer
* participants who express a refusal to provide informed consent

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size, determined by insights from a study by An J, which showcased a median 10-year ASCVD risk of 0.6% in a sizable sample of 414,260 young adults, has been rigorously calculated. To enhance the robustness of our study and account for potential observational bias and missing clinical characteristics, the initially identified sample size has been increased by a factor of 1.5. This adjustment ensures a more comprehensive representation, resulting in a final sample size of 3,513 individuals, specifically young and healthy participants. To accurately reflect the diverse population across Pakistan, stratification based on the 2017 census data will be employed, ensuring representation from all four provinces and optimizing the study's applicability and generalizability.
Sampling Method: Non-Probability Sample
Enrollment: 3513 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
10-year ASCVD risk Categorization | 3 Months
  Participants will be stratified into distinct 10-year ASCVD risk categories, including low risk (<5%), borderline risk (5% to <7.5%), intermediate risk (7.5% to <20%), or high risk (≥20%).
30-year ASCVD risk Categorization | 3 Months
  The 30-year ASCVD risk assessment will utilize the formula proposed by Pencina MJ, classifying participants based on their risk for "hard" and "general" CVD events.
Lifetime ASCVD risk evaluation | 3 Months
  The lifetime ASCVD risk evaluation will categorize individuals into risk groups, distinguishing between optimal, not optimal, elevated, and major risk factors, determined by specific risk criteria.
Genetic Risk Assessment of ApoB | 3 Months
  For Genetic Risk Assessment of ApoB, the study will compute the Genetic Risk Score (GRS) based on genotyping the APOB rs1042031 variant, following the methodology outlined by Shahid SU. The unweighted GRS for ApoB will be derived through an additive approach, assigning values of 0, 1, and 2 for protective homozygous, heterozygous, and risk homozygous genotypes, respectively. This resulting GRS for ApoB will range from 0 (indicating the absence of risk alleles) to 2 (both alleles identified as risk alleles for APOB rs1042031) in an individual.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Ashraf, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- Advanced Education Institute and Research Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mensah GA, Roth GA, Fuster V. The Global Burden of Cardiovascular Diseases and Risk Factors: 2020 and Beyond. J Am Coll Cardiol. 2019 Nov 19;74(20):2529-2532. doi: 10.1016/j.jacc.2019.10.009. No abstract available. PMID 31727292
- [Background] Connelly PJ, Azizi Z, Alipour P, Delles C, Pilote L, Raparelli V. The Importance of Gender to Understand Sex Differences in Cardiovascular Disease. Can J Cardiol. 2021 May;37(5):699-710. doi: 10.1016/j.cjca.2021.02.005. Epub 2021 Feb 13. PMID 33592281
- [Background] Wang T, Zhao Z, Yu X, Zeng T, Xu M, Xu Y, Hu R, Chen G, Su Q, Mu Y, Chen L, Tang X, Yan L, Qin G, Wan Q, Gao Z, Wang G, Shen F, Luo Z, Qin Y, Chen L, Huo Y, Li Q, Ye Z, Zhang Y, Liu C, Wang Y, Wu S, Yang T, Deng H, Zhao J, Xu Y, Li M, Chen Y, Wang S, Ning G, Bi Y, Shi L, Lu J, Wang W. Age-specific modifiable risk factor profiles for cardiovascular disease and all-cause mortality: a nationwide, population-based, prospective cohort study. Lancet Reg Health West Pac. 2021 Sep 26;17:100277. doi: 10.1016/j.lanwpc.2021.100277. eCollection 2021 Dec. PMID 35005664
- [Background] Zhao D. Epidemiological Features of Cardiovascular Disease in Asia. JACC Asia. 2021 Jun 15;1(1):1-13. doi: 10.1016/j.jacasi.2021.04.007. eCollection 2021 Jun. PMID 36338365
- [Background] Gheorghe A, Griffiths U, Murphy A, Legido-Quigley H, Lamptey P, Perel P. The economic burden of cardiovascular disease and hypertension in low- and middle-income countries: a systematic review. BMC Public Health. 2018 Aug 6;18(1):975. doi: 10.1186/s12889-018-5806-x. PMID 30081871
- [Background] Joseph P, Leong D, McKee M, Anand SS, Schwalm JD, Teo K, Mente A, Yusuf S. Reducing the Global Burden of Cardiovascular Disease, Part 1: The Epidemiology and Risk Factors. Circ Res. 2017 Sep 1;121(6):677-694. doi: 10.1161/CIRCRESAHA.117.308903. PMID 28860318
- [Background] Lu Y, Li SX, Liu Y, Rodriguez F, Watson KE, Dreyer RP, Khera R, Murugiah K, D'Onofrio G, Spatz ES, Nasir K, Masoudi FA, Krumholz HM. Sex-Specific Risk Factors Associated With First Acute Myocardial Infarction in Young Adults. JAMA Netw Open. 2022 May 2;5(5):e229953. doi: 10.1001/jamanetworkopen.2022.9953. PMID 35503221
- [Background] Cho KI, Shin ES, Ann SH, Garg S, Her AY, Kim JS, Han JH, Jeong MH; KAMIR Registry. Gender differences in risk factors and clinical outcomes in young patients with acute myocardial infarction. J Epidemiol Community Health. 2016 Nov;70(11):1057-1064. doi: 10.1136/jech-2015-207023. Epub 2016 May 4. PMID 27146351
- [Background] Batra MK, Rizvi NH, Sial JA, Saghir T, Karim M. Angiographic characteristics and in hospital outcome of young patients, age up to 40 versus more than 40 years undergoing primary percutaneous coronary intervention. J Pak Med Assoc. 2019 Sep;69(9):1308-1312. PMID 31511716
- [Background] Ullah W, Malik R, Bashir F, Khan M, Khan S, Alam M, Samad Z, Achirica MC, Virani SS, Hanif B. Comparison of Premature, Extremely Premature, and Older Adults With Coronary Artery Disease in Pakistan. JACC Asia. 2023 Jan 24;3(1):164-165. doi: 10.1016/j.jacasi.2022.10.002. eCollection 2023 Feb. No abstract available. PMID 36873748
- [Background] Studzinski K, Tomasik T, Krzyszton J, Jozwiak J, Windak A. Effect of using cardiovascular risk scoring in routine risk assessment in primary prevention of cardiovascular disease: an overview of systematic reviews. BMC Cardiovasc Disord. 2019 Jan 9;19(1):11. doi: 10.1186/s12872-018-0990-2. PMID 30626326
- [Background] Goff DC Jr, Lloyd-Jones DM, Bennett G, Coady S, D'Agostino RB, Gibbons R, Greenland P, Lackland DT, Levy D, O'Donnell CJ, Robinson JG, Schwartz JS, Shero ST, Smith SC Jr, Sorlie P, Stone NJ, Wilson PW, Jordan HS, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S49-73. doi: 10.1161/01.cir.0000437741.48606.98. Epub 2013 Nov 12. No abstract available. PMID 24222018
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] An J, Zhang Y, Zhou H, Zhou M, Safford MM, Muntner P, Moran AE, Reynolds K. Incidence of Atherosclerotic Cardiovascular Disease in Young Adults at Low Short-Term But High Long-Term Risk. J Am Coll Cardiol. 2023 Feb 21;81(7):623-632. doi: 10.1016/j.jacc.2022.11.051. PMID 36792277
- [Background] Lloyd-Jones DM, Braun LT, Ndumele CE, Smith SC Jr, Sperling LS, Virani SS, Blumenthal RS. Use of Risk Assessment Tools to Guide Decision-Making in the Primary Prevention of Atherosclerotic Cardiovascular Disease: A Special Report From the American Heart Association and American College of Cardiology. J Am Coll Cardiol. 2019 Jun 25;73(24):3153-3167. doi: 10.1016/j.jacc.2018.11.005. Epub 2018 Nov 10. PMID 30423392
- [Background] Lee CK, Liao CW, Meng SW, Wu WK, Chiang JY, Wu MS. Lipids and Lipoproteins in Health and Disease: Focus on Targeting Atherosclerosis. Biomedicines. 2021 Aug 9;9(8):985. doi: 10.3390/biomedicines9080985. PMID 34440189
- [Background] Mehta A, Shapiro MD. Apolipoproteins in vascular biology and atherosclerotic disease. Nat Rev Cardiol. 2022 Mar;19(3):168-179. doi: 10.1038/s41569-021-00613-5. Epub 2021 Oct 8. PMID 34625741
- [Background] Behbodikhah J, Ahmed S, Elyasi A, Kasselman LJ, De Leon J, Glass AD, Reiss AB. Apolipoprotein B and Cardiovascular Disease: Biomarker and Potential Therapeutic Target. Metabolites. 2021 Oct 8;11(10):690. doi: 10.3390/metabo11100690. PMID 34677405
- [Background] Sniderman AD, Thanassoulis G, Glavinovic T, Navar AM, Pencina M, Catapano A, Ference BA. Apolipoprotein B Particles and Cardiovascular Disease: A Narrative Review. JAMA Cardiol. 2019 Dec 1;4(12):1287-1295. doi: 10.1001/jamacardio.2019.3780. PMID 31642874
- [Background] Lawler PR, Akinkuolie AO, Ridker PM, Sniderman AD, Buring JE, Glynn RJ, Chasman DI, Mora S. Discordance between Circulating Atherogenic Cholesterol Mass and Lipoprotein Particle Concentration in Relation to Future Coronary Events in Women. Clin Chem. 2017 Apr;63(4):870-879. doi: 10.1373/clinchem.2016.264515. Epub 2017 Feb 7. PMID 28174174
- [Background] Welsh C, Celis-Morales CA, Brown R, Mackay DF, Lewsey J, Mark PB, Gray SR, Ferguson LD, Anderson JJ, Lyall DM, Cleland JG, Jhund PS, Gill JMR, Pell JP, Sattar N, Welsh P. Comparison of Conventional Lipoprotein Tests and Apolipoproteins in the Prediction of Cardiovascular Disease. Circulation. 2019 Aug 13;140(7):542-552. doi: 10.1161/CIRCULATIONAHA.119.041149. Epub 2019 Jun 20. PMID 31216866
- [Background] Visseren FLJ, Mach F, Smulders YM, Carballo D, Koskinas KC, Back M, Benetos A, Biffi A, Boavida JM, Capodanno D, Cosyns B, Crawford C, Davos CH, Desormais I, Di Angelantonio E, Franco OH, Halvorsen S, Hobbs FDR, Hollander M, Jankowska EA, Michal M, Sacco S, Sattar N, Tokgozoglu L, Tonstad S, Tsioufis KP, van Dis I, van Gelder IC, Wanner C, Williams B; ESC National Cardiac Societies; ESC Scientific Document Group. 2021 ESC Guidelines on cardiovascular disease prevention in clinical practice. Eur Heart J. 2021 Sep 7;42(34):3227-3337. doi: 10.1093/eurheartj/ehab484. No abstract available. PMID 34458905
- [Background] Pencina MJ, D'Agostino RB Sr, Larson MG, Massaro JM, Vasan RS. Predicting the 30-year risk of cardiovascular disease: the framingham heart study. Circulation. 2009 Jun 23;119(24):3078-84. doi: 10.1161/CIRCULATIONAHA.108.816694. Epub 2009 Jun 8. PMID 19506114
- [Background] Shahid SU, Shabana, Cooper JA, Beaney KE, Li K, Rehman A, Humphries SE. Genetic risk analysis of coronary artery disease in Pakistani subjects using a genetic risk score of 21 variants. Atherosclerosis. 2017 Mar;258:1-7. doi: 10.1016/j.atherosclerosis.2017.01.024. Epub 2017 Jan 22. PMID 28167353